CLINICAL TRIAL: NCT03109054
Title: Role of Endogenous Melatonin Level in Preoperative and Postoperative Anxiety in Bariatric Surgery Patients
Brief Title: Endogenous Melatonin Level and Pre- Postoperative Anxiety in Bariatric Surgery Patients.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Mehmet Ali Erdoğan, Associate Professor, M.D., Inonu University
Other Study IDs: MAE4
Record Dates: First submitted 2017-03-28; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Anxiety Disorders; Melatonin
Keywords: Melatonin; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Anxiety Level: The patients had low anxiety levels. Anxiety levels will determine with S-Anxiety TX-1 (State-Trait Anxiety Inventory Test:https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3879951/)
  Interventions: Diagnostic Test: State-Trait Anxiety Inventory Test
- High Anxiety Level: The patients had high anxiety levels. Anxiety levels will determine with S-Anxiety (State-Trait Anxiety Inventory Test: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3879951/)
  Interventions: Diagnostic Test: State-Trait Anxiety Inventory Test

INTERVENTIONS:
Diagnostic Test: State-Trait Anxiety Inventory Test — All patients will take a State-Trait Anxiety Inventory Test. After the test patients will enroll low or high anxiety level.
  Other Names: STAI FORM TX-1

SUMMARY:
Bariatric surgical procedures are associated with low short-term mortality and may be associated with long-term reductions in all-cause, cardiovascular, and cancer-related mortality. This surgeries are major surgeries include risk of mortality still.

Different level anxiety that can define as fear or worry can be seen in 60%-80% of patients scheduled surgery. Anxiety levels; may vary on age, gender, type of operation, previous experience of anesthesia and surgery and way of hospitalization. Preoperative anxiety affects negatively the surgery, the anesthesia and postoperative recovery.

Melatonin is a hormone secreted from the pineal gland. The circadian rhythm of melatonin changes according to age and it's production decreases with older ages. Melatonin is an antioxidant, antinociceptive, hypnotic, anticonvulsant, neuroprotective, anxiolytic, sedative, analgesic and has a preventive effect of delirium in intensive care. Irregularity of melatonin secretion causes a sleep irregularities, psychosis in intensive care unit and some behavioral disorder. It has been demonstrated that oral exogen administration of melatonin was effective on preoperative anxiety.

The aim of this study was to determine the relationship between endogenous melatonin levels and anxiety levels in patients with bariatric surgery.

DETAILED DESCRIPTION:
Bariatric surgical procedures, including gastric bypass, vertical sleeve gastrectomy, and biliopancreatic diversion, are the most effective and durable treatments for obesity. Bariatric surgery provides long-term benefit for patients with diabetes, fatty liver disease, and other metabolic disorders, through both weight loss-dependent and -independent mechanisms.

Bariatric surgery is associated with low short-term mortality and may be associated with long-term reductions in all-cause, cardiovascular, and cancer-related mortality. This surgeries are major surgeries include risk of mortality still.

Different level anxiety that can define as fear or worry can be seen in 60%-80% of patients scheduled surgery. Anxiety levels; may vary on age, gender, type of operation, previous experience of anesthesia and surgery and way of hospitalization. Preoperative anxiety affects negatively the surgery, the anesthesia and postoperative recovery. It may cause the pathophysiological response as hypertension and arrhythmia even refusal the surgery is planned. Also the anesthetic requirements and the risk "awareness" during the operation may increase. Patients with high level anxiety have more postoperative pain symptoms too. Therefore determination of the causes and prevention of anxiety is important.

Melatonin is a hormone secreted from the pineal gland, also known as the pineal gland. It's production is stimulated by darkness, independent of sleep, and is inhibited by exposure to light and proved endocrine rhythms. It shows a daily biorhythm. The circadian rhythm of melatonin changes according to age and it's production decreases with older ages. Melatonin level can be measured in the blood and in urine collected for 24 hours. Melatonin is an antioxidant, antinociceptive, hypnotic, anticonvulsant, neuroprotective, anxiolytic, sedative, analgesic and has a preventive effect of delirium in intensive care. Irregularity of melatonin secretion causes a sleep irregularities, psychosis in intensive care unit and some behavioral disorder. It has been demonstrated that oral exogen administration of melatonin was effective on preoperative anxiety.

The aim of this study was to determine the relationship between endogenous melatonin levels and anxiety levels in patients with bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologists (ASA) 3-4 status, aged between 18-65 years who are scheduled to undergo bariatric surgery.

Exclusion Criteria:

Patients with cardiovascular and pulmonary disease, those with ASA III-IV and propofol, fentanyl, remifentanil and rocuronium allergy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients of American Society of Anesthesiologists (ASA) 1-2 status, aged between 18-65 years who are scheduled to undergo bariatric surgery, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-05-15 (Estimated); Study Completion 2017-06-15 (Estimated)

PRIMARY OUTCOMES:
change in melatonin levels | preoperative and 24. hour after postoperative
  Melatonin is a hormone secreted from the pineal gland. It shows a daily biorhythm. The circadian rhythm of melatonin changes according to age and it's production decreases with older ages. Melatonin level can be measured in the blood and in urine collected for 24 hours.

SECONDARY OUTCOMES:
S-Anxiety (State-Trait Anxiety Inventory Test | preoperative and 24. hour after postoperative
  Anxiety levels; may vary on age, gender, type of operation, previous experience of anesthesia and surgery and way of hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu university, Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
no a plan

REFERENCES:
- [Result] Cardoso L, Rodrigues D, Gomes L, Carrilho F. Short- and long-term mortality after bariatric surgery: A systematic review and meta-analysis. Diabetes Obes Metab. 2017 Sep;19(9):1223-1232. doi: 10.1111/dom.12922. Epub 2017 May 31. PMID 28244626
- [Result] Hansen MV. Chronobiology, cognitive function and depressive symptoms in surgical patients. Dan Med J. 2014 Sep;61(9):B4914. PMID 25186550
- [Result] Edwards-Hampton SA, Madan A, Wedin S, Borckardt JJ, Crowley N, Byrne KT. A closer look at the nature of anxiety in weight loss surgery candidates. Int J Psychiatry Med. 2014;47(2):105-13. doi: 10.2190/PM.47.2.b. PMID 25084797